CLINICAL TRIAL: NCT03132064
Title: The Association Between Pre-operative Pain Psychology and Hypersensitivity With Poor Functional Outcome After Knee Replacement
Status: Suspended | Type: Observational
Why Stopped: COVID-19
Sponsor: University of Salford (Other)
Collaborators: Stockport NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Bodor Bin sheeha, Principal Investigator -PhD student at University of Salford, University of Salford
Other Study IDs: usalford- prospective
Record Dates: First submitted 2017-04-11; First posted 2017-04-27 (Actual); Last update posted 2020-05-27 (Actual); Status verified 2020-05

CONDITIONS: Outcome After Total Knee Arthroplasty
MeSH Terms: interventions — Arthroplasty, Replacement, Knee

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- post total knee arthroplasty: The measurements will made for patients before and after total knee arthroplasty to explore the improvements and possible correlation with preoperative pain psychology and hypersensitivity
  Interventions: Procedure: total knee arthroplasty

INTERVENTIONS:
Procedure: total knee arthroplasty — surgical repair for end stage of knee osteoarthritis.
  Other Names: total knee replacement surgery

SUMMARY:
To explore whether there are factors that help us to understand why some patient outcomes are not successful and identify prediction factors for progression. Assess central pain sensitisation and psychology pre- and post-surgery with reliable tools that explore prediction tools for good/poor progression and improve patient selection, patient preparation and timing for surgery.

The aim of this project is to explore the effects of pre-surgical central pain sensitisation on pain and function outcomes post-TKA. Central pain sensitisation will be assessed using pressure algometry and the Pain Catastrophizing Scale will be used to explore pain psychology. Functional outcomes post-TKA will be assessed using a commonly used scale for patients' self-reported outcomes (Oxford Knee Score), visual analogue scale, a star excursion balance test and four recommended patient performance-based tests.

DETAILED DESCRIPTION:
Knee osteoarthritis (OA) is a major cause of disability around the world; it is the most common chronic condition in primary care in the UK. By 2030 it is predicted to be the greatest cause of disability in the general population. An effective end-stage treatment for knee OA is knee-replacement surgery, which was first done in the 1970s and 1980s.

In England and Wales, the number of knee-replacement procedures recorded by the National Joint Registry in 2013 was 91,703, which represents an increase of 0.9 % over 2012. The data analysis by the National Joint Registry and the Office of National Statistics suggests that, by 2030, primary TKAs will increase by 117% from the 2012 level. Subsequently, TKA revision surgeries are expected to increase incrementally by 332%. There is a similar estimation of demand for revision TKA surgeries in the United States; by 2030, they are expected to rise by 601% from the 2005 level. The United States estimation of primary TKA is for growth of 673% from the 2005 level, which is similar to England and Wales's upper-limit projections.

Post-TKA, 75-85% of patients report satisfaction with surgery outcomes, while the remaining 15-25% are dissatisfied . Total knee arthroplasty's success has traditionally been evaluated from the surgeon's perspective, e.g. the presence of surgical complications or implant survival. This is gradually changing to involve the patient in measuring health outcomes and decision-making processes. Patient-reported outcome measures (PROMs) have evolved to explore patient perspectives by monitoring the quality of care in health organizations and conducting clinical trial outcomes.

Worldwide National Joint Registry summarise the common indication for TKA revision are; 29.8% due to aseptic loosening, 14.8% infection and 9.5% due to pain. Most prediction studies show that pain and psychology pre-operation may predict poor outcomes post-TKA. A systematic review by concludes that pain catastrophizing predicts chronic pain post-TKA. Pain catastrophizing is defined as a construct that reflects anxious preoccupation with pain, an inability to inhibit pain-related fears, amplification of the significance of pain vis-à-vis health implications, and a sense of helplessness regarding pain.

Chronic post-surgery pain is significantly associated with preoperational central sensitisation as in post-shoulder subacrominal decompression and hernia repair. Regarding post-TKA, a study by Lundblad et al. (2008) concluded that the preoperational hand electrical pain threshold significantly predicts pain outcomes one year post-TKA. The study explored the association between chronic pain post-TKA and preoperation widespread pain sensitisation using pressure algometry. Both study association without control the psychological confiding factor. The correlation with Western Ontario and McMaster Universities Osteoarthritis Index pain score (WOMAC) is questionable due to weakness of WOMAC with post TKA population such as low sensitivity of WOMAC's stiffness subscale reduces the overall standardized response mean and high ceiling effect Psychological pain thinking is assessed using the most widely used measuring scale: Pain Catastrophizing Scale (PCS). PCS assesses pain thinking in three dimensions: rumination ("I can't stop thinking about how much it hurts"), magnification ("I worry that something serious may happen") and helplessness ("It's awful and I feel that it overwhelms me").

The current study will investigate preoperational central sensitisation using pressure algometry, in addition to the Pain Catastrophizing Scale (PCS), to explore psychological factors. There may be some correlation between preoperational central sensitisation and post-TKA outcomes such as pain and functional improvements.

To the best of our knowledge, no previous study has explored central sensitisation using pressure algometry and the Pain Catastrophizing Scale and possible correlation with its effects on pain and function recovery post-TKA. Pain and function can be accurately assessed before and after TKA using visual analogue scale, Oxford Knee Score, balance and performance functional tests. No previous study has correlated preoperational central sensitisation and pain psychology post-TKA on the Oxford Knee Scale as commonly used patients' self-reported outcome measures.

Thus, the study may explore accurate and objective prediction factors of post-total-knee arthroplasty progression. Potentially, reliable outcome prediction could, however, improve patient selection for surgery, as appropriate timing for surgery depends on patient symptoms and efficient patient preparation for surgery if it is to be cost-effective. Accurate preoperative prediction is crucial to minimize the potential for unrealistic expectations.

ELIGIBILITY:
Inclusion Criteria:

* All patients scheduled for elective primary unilateral total knee arthroplasty for end-stage knee osteoarthritis with stable and controlled medical condition

Exclusion Criteria:

Potential research participants were excluded from the study if ;

* The patients schedule for bilateral knee arthroplasty or unilateral knee revision surgery.
* The patient cannot read and understand English language.
* Their function limited due to other musculoskeletal involvements other than unilateral knee osteoarthritis.
* Diagnosed with uncontrolled diabetes mellitus or blood pressure.
* Diagnosed with any neurologic disorders such as stroke, Parkinson disease or multiple sclerosis.
* morbid obese patients their body mass index BMI greater than 40.
* Advance osteoporosis or other unstable chronic disease.
* Diagnosed with peripheral vascular diseases or uncontrolled cardiac diseases.
* The participant will excluded post-surgery if they develop any surgical complication such as deep vein thrombosis, uncontrolled infection, or fracture

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The present study is a prospective randomised 6 months follow-up. All patients scheduled for elective primary unilateral total knee arthroplasty for end-stage knee osteoarthritis with stable and controlled medical condition will asked for participation in preadmission orthopaedics clinic visit at Stepping Hill Hospital. The information sheet will give to all participants agreed to participate to clarify the objective of study (Appendix 1). Before commencement, patients will sign a consent form (Appendix 2) and have the right to clarify any enquiry regarding the study with the researcher. The patient's participation will not affect the quality of service, all patients will received conventional orthopaedic care and a standard amount of physiotherapy according to hospital protocols.
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2020-09-12 (Estimated); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Changes in Pain Catastrophizing Scale (PCS) | before surgery and 6 months after
  Catastrophizing contributes to heightened levels of pain, emotional distress, chronic pain and disability (Forsythe, Dunbar, Hennigar, Sullivan, & Gross, 2008).
  The PCS has 13 items and can be completed and scored in less than 5 minutes. It reflects past painful experiences and indicates the degree to which patients experience each of 13 thoughts or feelings when in pain. It has 5-point scales with end points (0) not at all and (4) all the time. Between the 50th and 75th percentiles of PCS score, patients are considered at moderate risk and at more than the 75th percentile they are consider at high risk for developing chronicity. It is a reliable and valid catastrophizing measure, it shows excellent internal consistency, total score coefficient alphas = .87-.93 and significant correlation with the Inventory of Negative Thoughts in Response to Pain scale and general psychological disturbance (MASQGeneral Disturbance) scale (Osman et al., 1997; Sullivan & et al., 1995) (Appendix 3).
Changes in Central Sensitisation using pressure algometry | before surgery and 6 months after
  Pressure will be applied using a handheld pressure algometer (Algometer Type II, Somedic AB, Sweden) at a rate of 30 kPa/s perpendicular to the skin with a 1 cm² probe. The pressure pain threshold will be estimated by instructing participants to say 'stop' when the sensation of pressure becomes the first sensation of pain (Arendt-Nielsen et al., 2010; Lunn, Kristensen, Gaarn-Larsen, & Kehlet, 2012; Skou et al., 2013). Pressure will be applied to the medial side of the operated knee and the volar surface of the same side forearm. These two body sites are chosen because they represent painful areas in knee OA patients and may provide evidence of widespread pain sensitisation (forearm) and localised pain sensitisation (knee) (Wylde, Palmer, Learmonth, & Dieppe, 2011; Wylde et al., 2013). The site for knee pressure will be at 3 cm medial to the midpoint on the medial edge of the index patella

SECONDARY OUTCOMES:
Changes in Oxford Knee Score (OKS) | before surgery and 6 months after
  A final version of a 12-item questionnaire was developed to assess patients post-TKA after interviews with patients undergoing joint replacement and a multiple drafting process to identify their experiences and problems post-TKA since 1998 (Appendix 4).
  OKS is a valid, reliable and responsive assessment tool for the period post-TKA, it has advantages over the Western Ontario and McMaster Universities Osteoarthritis Index - Knee Injury and Osteoarthritis Outcome Score, as it simple and short. As a PROM's main concern is to explore outcomes from the patient's perspective, OKS has the advantage of offering clear MIDC values for all types of study and is designed to ensure that results are recognized by patients, in addition to statistical differences, and this may improve the power calculation (Beard et al., 2015; Clement, MacDonald, Patton, & Burnett, 2015; Clement, MacDonald, & Simpson, 2014; Dawson, Fitzpatrick, Murray, & Carr, 1998)
Changes in pain visual analogue scale (VAS); | before surgery and 6 months after
  The pain visual analogue scale will used to assess the pain before and after the surgery. The scale consist of a 100 mm long horizontal line ranging from no pain to intolerable pain (Appendix 4). Patients will instruct to mark the line at the point matched their pain. The assessor will measure with ruler the millimetres and converted to points (0 points no pain to 100 points intolerable pain) (Bullens, van Loon, de Waal Malefijt, Laan, & Veth, 2001).
Changes in Assessment of Performance based measurements (30 s chair-stand test) | before surgery and 6 months after
  Based in published protocol, the chair with 17 inches (45cm) height with starting position will be sitting with arm cross the chest. The patients will instruct to stand then sit with good buttock placement, back support, hand on arm rest and foot placements then stand again as fast and safe as they can. The assessor will count the number of complete chair stand within the 30 second. The mean of two trail will use for analysis (Gill & McBurney, 2008; Unver, Kalkan, Yuksel, Kahraman, & Karatosun, 2015).
Changes in stair-climb test | before surgery and 6 months after
  The assessor will measure the time required using timed stopwatch within one hundredth of second using one handrail if required to ascend and descend flight of twelve 18-cm-high steps and 28 cm depth. The patients will instruct to ascend and descend the stairs as quickly, safe and comfortable they can. The mean of two trail will use for analysis (Mizner et al., 2011).
Changes in Timed up-and-go test | before surgery and 6 months after
  According to published protocol the test procedure will be as following based on used timed stopwatch within one hundredth of second, standard height chair of 45cm with arm rest will placed on an outdoor level footpath and a line 3 meters from the chair will draw. The patients will instruct to rise from chair using the arms if required, walk for 3 meter until the line mark then turn back to sit on the chair as quickly, safe and comfortable they can. The assessor commenced timing as the patient leaned forward to stand up, and stop when the patient hips made contact with the seat to sit down. Average of 3 performance will analysis (Ko, Naylor, Harris, Crosbie, & Yeo, 2013; Mizner et al., 2011; Podsiadlo & Richardson, 1991).
Changes in Six minute walk test | before surgery and 6 months after
  Based on the test published guideline the test will measure how far the patients can walk in 6 minute in level surface, 25 meter footpath. The patient can use the assistive device if required, take rest if need with standardized encouragement after each minute. The assessor will ask the patient to stop at 6 minute. One test will be perform to avoid fatigue ("ATS Statement," 2002; Ko et al., 2013; Mizner et al., 2011).
Changes in Balance Test | before surgery and 6 months after
  Balance will be assessed using the simple Star Excursion Balance Test, which is considered to be a reliable, valid dynamic test to identify dynamic balance deficits in patients with lower extremity conditions. The assessor will measure the reach distance in each direction in centimetres and then normalise the average of the three trials to leg length. Limb length will be measured while lying in a supine position from anterior superior iliac spine to the centre of the ipsilateral medial malleolus. Reach distances will be normalised to limb length by calculating the maximum reach distance (%MAXD) using the formula (excursion distance/limb length) ×100 (Coughlan, Fullam, Delahunt, Gissane, & Caulfield, 2012; Fullam et al., 2014; Robinson & Gribble, 2008).
Changes in Physical activity | before surgery and 6 months after
  measurements will be made using an activPAL activity monitor (PAL Technologies, Glasgow, UK) as this proven accelerometer provides objective quantification of free-living physical activity without any modification (Dahlgren, Carlsson, Moorhead, Hager-Ross, & McDonough, 2010; Schmalzried et al., 1998). It is suitable as it light in weight (20g), includes an inclinometer and is small in size (53 x 35 x 7 mm) Figure 3. The device is worn by patient's mid-thigh, secured by non-allergic waterproof adhesive tape under their clothes, for 7-10 days before surgery and 6 months after. Clear written and verbal instructions will be given to patients as they have to wear it all day and all night except, when bathing or swimming (they can take a shower with it on).

CONTACTS AND LOCATIONS:
Locations (1):
- Stockport NHS Foundation Trust, Stockport, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Arendt-Nielsen L, Nie H, Laursen MB, Laursen BS, Madeleine P, Simonsen OH, Graven-Nielsen T. Sensitization in patients with painful knee osteoarthritis. Pain. 2010 Jun;149(3):573-581. doi: 10.1016/j.pain.2010.04.003. Epub 2010 Apr 24. PMID 20418016
- [Background] Bade MJ, Wolfe P, Zeni JA, Stevens-Lapsley JE, Snyder-Mackler L. Predicting poor physical performance after total knee arthroplasty. J Orthop Res. 2012 Nov;30(11):1805-10. doi: 10.1002/jor.22140. Epub 2012 Apr 26. PMID 22539338
- [Background] Beard DJ, Harris K, Dawson J, Doll H, Murray DW, Carr AJ, Price AJ. Meaningful changes for the Oxford hip and knee scores after joint replacement surgery. J Clin Epidemiol. 2015 Jan;68(1):73-9. doi: 10.1016/j.jclinepi.2014.08.009. Epub 2014 Oct 31. PMID 25441700
- [Background] Burns LC, Ritvo SE, Ferguson MK, Clarke H, Seltzer Z, Katz J. Pain catastrophizing as a risk factor for chronic pain after total knee arthroplasty: a systematic review. J Pain Res. 2015 Jan 5;8:21-32. doi: 10.2147/JPR.S64730. eCollection 2015. PMID 25609995
- [Background] Clement ND, MacDonald D, Patton JT, Burnett R. Post-operative Oxford knee score can be used to indicate whether patient expectations have been achieved after primary total knee arthroplasty. Knee Surg Sports Traumatol Arthrosc. 2015 Jun;23(6):1578-90. doi: 10.1007/s00167-014-2865-0. Epub 2014 Feb 1. PMID 24488224
- [Background] Clement ND, MacDonald D, Simpson AH. The minimal clinically important difference in the Oxford knee score and Short Form 12 score after total knee arthroplasty. Knee Surg Sports Traumatol Arthrosc. 2014 Aug;22(8):1933-9. doi: 10.1007/s00167-013-2776-5. Epub 2013 Nov 20. PMID 24253376
- [Background] Coughlan GF, Fullam K, Delahunt E, Gissane C, Caulfield BM. A comparison between performance on selected directions of the star excursion balance test and the Y balance test. J Athl Train. 2012 Jul-Aug;47(4):366-71. doi: 10.4085/1062-6050-47.4.03. PMID 22889651
- [Background] Dawson J, Fitzpatrick R, Murray D, Carr A. Questionnaire on the perceptions of patients about total knee replacement. J Bone Joint Surg Br. 1998 Jan;80(1):63-9. doi: 10.1302/0301-620x.80b1.7859. PMID 9460955
- [Background] Forsythe ME, Dunbar MJ, Hennigar AW, Sullivan MJ, Gross M. Prospective relation between catastrophizing and residual pain following knee arthroplasty: two-year follow-up. Pain Res Manag. 2008 Jul-Aug;13(4):335-41. doi: 10.1155/2008/730951. PMID 18719716
- [Background] Fullam K, Caulfield B, Coughlan GF, Delahunt E. Kinematic analysis of selected reach directions of the Star Excursion Balance Test compared with the Y-Balance Test. J Sport Rehabil. 2014 Feb;23(1):27-35. doi: 10.1123/jsr.2012-0114. Epub 2013 Aug 12. PMID 23945793
- [Background] Gandek B. Measurement properties of the Western Ontario and McMaster Universities Osteoarthritis Index: a systematic review. Arthritis Care Res (Hoboken). 2015 Feb;67(2):216-29. doi: 10.1002/acr.22415. PMID 25048451
- [Background] Giesinger K, Hamilton DF, Jost B, Holzner B, Giesinger JM. Comparative responsiveness of outcome measures for total knee arthroplasty. Osteoarthritis Cartilage. 2014 Feb;22(2):184-9. doi: 10.1016/j.joca.2013.11.001. Epub 2013 Nov 18. PMID 24262431
- [Background] Graven-Nielsen T, Wodehouse T, Langford RM, Arendt-Nielsen L, Kidd BL. Normalization of widespread hyperesthesia and facilitated spatial summation of deep-tissue pain in knee osteoarthritis patients after knee replacement. Arthritis Rheum. 2012 Sep;64(9):2907-16. doi: 10.1002/art.34466. PMID 22421811
- [Background] Gribble PA, Hertel J, Plisky P. Using the Star Excursion Balance Test to assess dynamic postural-control deficits and outcomes in lower extremity injury: a literature and systematic review. J Athl Train. 2012 May-Jun;47(3):339-57. doi: 10.4085/1062-6050-47.3.08. PMID 22892416
- [Background] Hertel J, Braham RA, Hale SA, Olmsted-Kramer LC. Simplifying the star excursion balance test: analyses of subjects with and without chronic ankle instability. J Orthop Sports Phys Ther. 2006 Mar;36(3):131-7. doi: 10.2519/jospt.2006.36.3.131. PMID 16596889
- [Background] Khan M, Osman K, Green G, Haddad FS. The epidemiology of failure in total knee arthroplasty: avoiding your next revision. Bone Joint J. 2016 Jan;98-B(1 Suppl A):105-12. doi: 10.1302/0301-620X.98B1.36293. PMID 26733654
- [Background] Lundblad H, Kreicbergs A, Jansson KA. Prediction of persistent pain after total knee replacement for osteoarthritis. J Bone Joint Surg Br. 2008 Feb;90(2):166-71. doi: 10.1302/0301-620X.90B2.19640. PMID 18256082
- [Background] Lungu E, Desmeules F, Dionne CE, Belzile EL, Vendittoli PA. Prediction of poor outcomes six months following total knee arthroplasty in patients awaiting surgery. BMC Musculoskelet Disord. 2014 Sep 8;15:299. doi: 10.1186/1471-2474-15-299. PMID 25201448
- [Background] Lunn TH, Kristensen BB, Gaarn-Larsen L, Kehlet H. Possible effects of mobilisation on acute post-operative pain and nociceptive function after total knee arthroplasty. Acta Anaesthesiol Scand. 2012 Nov;56(10):1234-40. doi: 10.1111/j.1399-6576.2012.02744.x. Epub 2012 Aug 10. PMID 22881199
- [Background] Osman A, Barrios FX, Kopper BA, Hauptmann W, Jones J, O'Neill E. Factor structure, reliability, and validity of the Pain Catastrophizing Scale. J Behav Med. 1997 Dec;20(6):589-605. doi: 10.1023/a:1025570508954. PMID 9429990
- [Background] Robinson RH, Gribble PA. Support for a reduction in the number of trials needed for the star excursion balance test. Arch Phys Med Rehabil. 2008 Feb;89(2):364-70. doi: 10.1016/j.apmr.2007.08.139. PMID 18226664
- [Background] Skou ST, Graven-Nielsen T, Rasmussen S, Simonsen OH, Laursen MB, Arendt-Nielsen L. Widespread sensitization in patients with chronic pain after revision total knee arthroplasty. Pain. 2013 Sep;154(9):1588-1594. doi: 10.1016/j.pain.2013.04.033. Epub 2013 Apr 20. PMID 23707268
- [Background] Sullivan, M. J. L., & et al. (1995). The Pain Catastrophizing Scale: Development and Validation. Psychological Assessment, 7(4), 524-532.
- [Background] Terwee CB, Bot SD, de Boer MR, van der Windt DA, Knol DL, Dekker J, Bouter LM, de Vet HC. Quality criteria were proposed for measurement properties of health status questionnaires. J Clin Epidemiol. 2007 Jan;60(1):34-42. doi: 10.1016/j.jclinepi.2006.03.012. Epub 2006 Aug 24. PMID 17161752
- [Background] Wylde V, Palmer S, Learmonth ID, Dieppe P. Test-retest reliability of Quantitative Sensory Testing in knee osteoarthritis and healthy participants. Osteoarthritis Cartilage. 2011 Jun;19(6):655-8. doi: 10.1016/j.joca.2011.02.009. Epub 2011 Feb 15. PMID 21329759
- [Background] Wylde V, Palmer S, Learmonth ID, Dieppe P. The association between pre-operative pain sensitisation and chronic pain after knee replacement: an exploratory study. Osteoarthritis Cartilage. 2013 Sep;21(9):1253-6. doi: 10.1016/j.joca.2013.05.008. PMID 23973138